CLINICAL TRIAL: NCT00457652
Title: Does Caffeine Reduce Rosuvastatin-Induced Protection Against Ischemia-Reperfusion Injury?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G Rongen, dept Pharmacology toxicology UMCN
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Rosuva01
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Ischemia Reperfusion Injury
Keywords: Rosuvastatin; Caffeine; Ischemia; Reperfusion
MeSH Terms: conditions — Reperfusion Injury; Ischemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 7 day treatment rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Placebo Comparator): 7 day treatment placebo
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — 7 day treatment rosuvastatin 20mg

SUMMARY:
Does caffeine reduce rosuvastatin induced protection against ischemia reperfusion injury?

DETAILED DESCRIPTION:
Rosuvastatin is a proven cholesterol lowering medicine, which hereby is assumed to achieve a reduction in cardiovascular events. Apart from it's cholesterol lowering action, rosuvastatin may also increase tolerance against ischemia-reperfusion injury. In dogs rosuvastatin increases the endogenous concentration of adenosine, by enhancing the activity of the enzyme ecto-5'-nucleotidase, which converts adenosine monophosphate into adenosine. We hypothesize that rosuvastatin increases tolerance against ischemia-reperfusion injury by induction of ecto-5'-nucleotidase and thereby increasing adenosine activity. This protective effect of rosuvastatin can be abrogated by using the adenosine receptor antagonist caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Male
* age between 18-50 yrs
* signed informed consent

Exclusion Criteria:

* Cardiovascular disease
* Hypertension (systole > 140 mmHg, diastole > 90 mmHg)
* Hypercholesterolemia (fasting total cholesterol > 6,0 mmol/l)
* Drug abuse
* Concomitant medication use
* Inability to perform the ischemic isometric muscle contraction
* Diabetes Mellitus (fasting glucose > 7.0 mmol/L or random glucose > 11.0 mmol/L)
* Alanine-Amino-Transferase (ALAT) >90U/L (more than twice the upper level of the normal range)
* Creatinine Kinase (CK) >340U/L (more than twice the upper level of the normal range)
* Participation in any trial concerning medicinal products during the last 60 days prior to this study.
* Participation in clinical trial involving

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The targeting of Technetium 99 labeled Annexin A5 is recorded with a gamma camera as a endpoint measure of ischemia-reperfusion damage. | 60 and 240 minutes after ischemic exercise

SECONDARY OUTCOMES:
Workload (product of 50% of the maximum forearm force and duration of the ischemic exercise) | during 10 minutes of ischemic exercise
The effect of one-week treatment of rosuvastatin 20mg once daily on lipid spectrum. | before and after 7day treatment
The caffeine serum concentration after 24 hour abstinence . | morning after 24 hours abstinence of caffeine

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, Phd, Principal Investigator — UMCN st. Radboud
Locations (1):
- UMCN st.Radboud, Nijmegen, Netherlands

REFERENCES:
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546
- [Derived] Meijer P, Oyen WJ, Dekker D, van den Broek PH, Wouters CW, Boerman OC, Scheffer GJ, Smits P, Rongen GA. Rosuvastatin increases extracellular adenosine formation in humans in vivo: a new perspective on cardiovascular protection. Arterioscler Thromb Vasc Biol. 2009 Jun;29(6):963-8. doi: 10.1161/ATVBAHA.108.179622. Epub 2009 Apr 9. PMID 19359665